CLINICAL TRIAL: NCT00361179
Title: An Extension, Observational Protocol to Evaluate the Long Term Effects of Peginterferon Alfa-2a Plus Ribavirin for Chronic Hepatitis C/B Co-Infection and Chronic Hepatitis C in the Original Study ML17862
Brief Title: Long Term Effects of Peginterferon Alfa-2a Plus Ribavirin for Chronic Hepatitis C/B Co-Infection and Chronic Hepatitis C
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Hoffmann-La Roche (Industry)
Other Study IDs: 9561706020
Record Dates: First submitted 2006-08-04; First posted 2006-08-07 (Estimated); Last update posted 2006-08-07 (Estimated); Status verified 2006-08

CONDITIONS: Coinfection With Hepatitis B Virus and Hepatitis C Virus; Monoinfection With Hepatitis C Virus
Keywords: Observation; Post-treatment
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Chronic hepatitis C may relapse in simple chronic hepatitis C patients who initially obtained sustained virologic responses. Although the HCV SVR could be maintained in around 90%, the remaining 10% of these patients may develop hepatitis C relapse during follow-up. Therefore, it is important to follow up the long-term of these patients with dual chronic hepatitis B and C.

From another aspect, for the treatment of chronic hepatitis B, the virologic and serologic responses may also not be durable. Alternatively, previous studies suggested that the therapeutic efficacy might not be seen in the study period, and incremental response might occur during long-term follow-up. Therefore it is also important to clarify the long-term outcome of treatment in this dually infected population.

Evaluation of the long term effects of treatment with peginterferon alfa-2a plus ribavirin for patients with chronic hepatitis C/ hepatitis B co-Infection and chronic hepatitis C in the original study ML17862 is important. This present protocol is thus to assess whether the HCV SVR is sustained and to assess the durability of the HBV virologic and serologic responses or any incremental response during a 5-year follow-up period, including six months after end of the therapy in the original study and an additional 4 and half years in this project (5 years overall follow-up after the end of treatment). Specifically, we wish to assess the (1) sustained virologic response (SVR) of HCV in both populations, (2) incidence of HBsAg loss and HBsAg seroconversion (HBsAg loss and appearance of anti-HBs) in dually infected population, (3) ALT normalization or flare off-treatment during both populations, (4) reductions of HCV RNA from the original baseline levels in the two patient populations, and (5) reduction of serum HBV DNA off-treatment in the dually infected population.

DETAILED DESCRIPTION:
Pegylated IFNs (such as PEG-IFN alfa-2a, PEGASYS®) have been shown to possess a superior efficacy and convenience to conventional IFNs, either alone or in combination with RBV in patients with chronic hepatitis C only [Zeuzem et al, 2000; Heathcote et al, 2000; Fried et al, 2002; Hadziyannis et al, EASL 2002]. For patients with chronic hepatitis B, pilot study also revealed that the biochemical and virologic responses were better in HBeAg-positive patients receiving pegylated IFN than those receiving conventional IFN [24-week post-treatment combined virologic, HBeAg loss, and ALT normalization rate: 28% vs. 12%; Lai et al, APSAL 2002].

The efficacy using a 24-week combination therapy in the sustained clearance of serum HCV RNA is equivalent to that using a 48-week combination therapy in patients with HCV genotype non-1 [Hadziyannis et al, EASL 2002]. A 48-week course of pegylated IFN and RBV combination therapy, in contrast, has been shown to yield a better efficacy in the sustained clearance of serum HCV RNA in patients with HCV genotype 1 than a 24-week combination therapy in western countries [SVR: 40~51% vs. 29~41%, Table 1, Hadziyannis et al, EASL 2002; Poynard et al, 1998]. Based on these findings, NIH Consensus Statement suggests that patients with genotype 1 need 48 weeks of combination treatment and standard doses of RBV [NIH 2002]. Previous study revealed that a 12-week RBV therapy was not effective for patients with chronic hepatitis B [Kakumu et al, 1993]. Therefore, in this proposal, the treatment duration will be 24 weeks for HCV genotype 2/3, and will be 48 weeks for HCV genotype 1, in patients with monoinfected chronic hepatitis C and dual chronic hepatitis C and B.

Increased RBV dosage has been considered as a contributory factor to the better efficacy in some previous studies. Recent studies suggested that using RBV 800 mg daily is adequate to treatment HCV genotype non-1 but standard dosage of RBV is required to treatment HCV genotype 1 [NIH 2002]. We follow the recommendations and use RBV 800 mg daily for HCV genotype non-1, both in dually infected patients and in monoinfected chronic hepatitis C patients. RBV with 1000-1200 mg daily will be used for HCV genotype 1 according the body weight of the patient, both in dually infected patients and in monoinfected chronic hepatitis C patients.

Previous studies suggested that chronic hepatitis C may relapse in simple chronic hepatitis C patients who initially obtained sustained virologic responses at 6 months after end of the treatment [Chemello et al, 1996; Marcellin et al, 1997]. Although the HCV SVR could be maintained in around 90%, the remaining 10% of these patients may develop hepatitis C relapse during follow-up. Chemello et al followed up 107 patients with chronic hepatitis C who maintained normal aminotransferase levels as long as 12 months after interferon-alpha therapy [Chemello et al, 1996]. Hepatitis C virus RNA was detected in 27 (25%) patients with sustained biochemical response; 80 (75%) patients were negative for HCV RNA. Patients positive for HCV RNA were older (P < 0.001), had received a smaller interferon-alpha dose (P = 0.02), and were more frequently infected with HCV genotype 2 (P < 0.01). Liver histologic findings were active in 57% of patients positive for HCV RNA, despite normal alanine aminotransferase levels, compared with only 12% of patients who were negative for HCV RNA (P = 0.01). The estimated probability of hepatitis relapse by 4 years after therapy was 53% in viremic patients and 0% in patients negative for HCV RNA (P < 0.001). Marcellin et al followed up 80 patients who had chronic hepatitis C and received interferon-alpha therapy [Marcellin et al, 1997]. The 80 patients had follow-up 1 to 7.6 years (mean +/- SD, 4.0 +/- 2.0 years) after interferon-alpha treatment. The follow-up period was 1, 2, 3, 4, 5, 6, and more than 6 years in 11, 13, 14, 18, 10, 12, and 2 patients, respectively, after the end of therapy. During the entire follow-up period, 93% (95% CI, 84% to 97%) of patients had persistently normal serum ALT levels. Serum HCV RNA remained undetectable in 96% (CI, 89% to 99%) of patients. A comparison of liver histologic findings before and 1 to 6.2 years after interferon-alpha treatment showed a clear improvement in 94% (CI, 83% to 99%) of patients. In 62% of patients, the last biopsy done showed normal or nearly normal histologic findings. Liver HCV RNA was detectable before treatment in all 13 patients tested and was undetectable 1 to 5 years after treatment in all 27 patients tested. They thus concluded that in patients with chronic hepatitis C who have persistently normal serum ALT levels and no detectable serum HCV RNA 6 months after interferon-alpha therapy, long-term sustained biochemical and virologic response is generally seen. Similar finding was noted in one reported case with dual chronic hepatitis B and C [Yalcin et al, 2003]. To be noted, this dually infected patient had reactivation of hepatitis B accompanied by severe flare of hepatitis activity during treatment and had relapse of hepatitis C after end of the treatment. Therefore, it is important to follow up the long-term of these patients with dual chronic hepatitis B and C.

From another aspect, for the treatment of chronic hepatitis B, the virologic and serologic responses may also not be durable [Liaw et al, 2005; Lok et al, 2004; Hadziyannis et al, 2003; Janssen et al, 2005]. Alternatively, previous studies suggested that the therapeutic efficacy might not be seen in the study period, and incremental response might occur during long-term follow-up as learned from previous experiences of using antiviral agents including interferon for the treatment of chronic hepatitis B [Saruc et al, 2003; Carreno et al, 2001]. Therefore it is also important to clarify the long-term outcome of treatment in this dually infected population.

This present protocol is thus to assess whether the HCV SVR is sustained and to assess the durability of the HBV virologic and serologic responses or any incremental response during a 5-year follow-up period, including six months after end of the therapy in the original study and an additional 4 and half years in this project (5 years overall follow-up after the end of treatment). Specifically, we wish to assess the (1) sustained virologic response (SVR) of HCV in both populations, (2) incidence of HBsAg loss and HBsAg seroconversion (HBsAg loss and appearance of anti-HBs) in dually infected population, (3) ALT normalization or flare off-treatment during both populations, (4) reductions of HCV RNA from the original baseline levels in the two patient populations, and (5) reduction of serum HBV DNA off-treatment in the dually infected population.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were randomized, treated and returned for follow up in the ML17862 protocol will be eligible for inclusion in this protocol

Exclusion Criteria:

* Patients unwilling to provide informed consent or abide by the requirements of the study.
* Patients who have already initiated anti-HCV or HBV treatment, approved or investigational since completion of the original protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320
Dates: Start 2006-05; Study Completion 2011-12

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Jer Chen, M.D.; Ph.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- Pei-Jer Chen, Taipei City, Taiwan, China

REFERENCES:
- [Derived] Liu CJ, Chuang WL, Lee CM, Yu ML, Lu SN, Wu SS, Liao LY, Chen CL, Kuo HT, Chao YC, Tung SY, Yang SS, Kao JH, Liu CH, Su WW, Lin CL, Jeng YM, Chen PJ, Chen DS. Peginterferon alfa-2a plus ribavirin for the treatment of dual chronic infection with hepatitis B and C viruses. Gastroenterology. 2009 Feb;136(2):496-504.e3. doi: 10.1053/j.gastro.2008.10.049. Epub 2008 Oct 29. PMID 19084016